CLINICAL TRIAL: NCT03265548
Title: Comparison Between Direct Laryngoscopy and Video Laryngoscopy for Neonatal Intubation. Confidence of Staff and Number of Attempts to Successful Intubation
Brief Title: Video Laryngoscopy in Newborn Babies V1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Derriford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16/SW/0013
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (No Intervention): Usual Direct view laryngoscopy
- Intervention (Experimental): Video laryngoscopy
  Interventions: Device: Video Laryngoscope

INTERVENTIONS:
Device: Video Laryngoscope — The use of video laryngoscopy
  Arms: Intervention

SUMMARY:
Our research questions are

1. Will the use of a video laryngoscope lead to decreased attempts
2. Does this result in more successful intubations and greater confidence in the supervisor and the team that a successful intubation has been performed.

DETAILED DESCRIPTION:
Neonatal intubation is a technically difficult, but essential, skill to learn, involving passing a plastic tube through the vocal cords, into the trachea. Current practice involves using a laryngoscope to directly visualise the cords, however this technique does not allow the supervisor to witness the tube passing through the cords. Video laryngoscopes have a camera at the distal end of the blade, allowing an 85% viewing angle as opposed to 15% that is seen with direct view. In addition, the image is projected onto a screen, allowing all members of the team to visualise the intubation and therefore provide real time guidance as well as increased confidence in the outcome of the attempt. Video laryngoscopes are used in neonates in other specialities, for example Ear Nose and throat or respiratory physicians, and are becoming routinely used by neonatologists. The research questions are whether using a video laryngoscope will lead to decreased attempts, which in turn will potentially result in more successful intubations and greater confidence in the supervisor and the team that a successful intubation has been performed.

The aim is to recruit 40 babies and randomly allocate the participant to either direct laryngoscopy or video laryngoscopy for elective intubations. Number of attempts to successful intubation would be recorded, in addition to confidence of supervisor and the team regarding the outcome of the attempt.

ELIGIBILITY:
Inclusion Criteria:

* Any baby requiring intubation on a neonatal unit

Exclusion Criteria:

* Infants will not be recruited if they are in extremis requiring immediate intubation by a senior experienced operator who will use his/her own preferred method. Infants who will be intubated nasally will not be included as this technique is not usually taught to registrars.

Any baby with a congenital airway malformation will not be included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of attempts to successful intubation | Each attempt is defined by the need to stop the attempt and give non-invasive support. A maximum of 3 attempts per trainee. The eligible participant is any baby on NNU who requires intubation
  How many attempts before successful intubation
Team confidence around tube placement at the time of tube placement | immediately after the intubation
  Continuous line to score the confidence of the individuals in the team

CONTACTS AND LOCATIONS:
Overall Officials: Bartle Dr David, MBChB, Principal Investigator — Consultant at Hospital
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No